CLINICAL TRIAL: NCT06299800
Title: Type 2 Diabetes Mellitus and Cancer: Phenotyping of Patients at a Third-level Diabetes Centre
Brief Title: Phenotyping Patients With Type 2 Diabetes Mellitus and Cancer
Acronym: TCPT2023
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE385/2023
Record Dates: First submitted 2024-02-13; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2; Cancer
Keywords: cancer; diabetes mellitus type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetes mellitus type 2 and cancer: 779 patients with cancer and diagnosis of type 2 diabetes mellitus diagnosed between 1990 and 2010
  Interventions: Other: phenotyping of patients followed at a third-level diabetes centre with cancer

INTERVENTIONS:
Other: phenotyping of patients followed at a third-level diabetes centre with cancer — Collection of the following data for each patient enrolled, where possible:
  * Gender and age;
  * Smoking habits and alcohol consumption (units per day);
  * Weight and body mass index (BMI) at first (T0) and last visit (T1);
  * Given by the diagnosis of type 2 diabetes mellitus;
  * Treatment of type 2 diabetes at T0 and T1;
  * Levels of glycated hemoglobin (hba1c) at T0 and T1, mean hba1c and mean fasting blood sugar;
  * Creatinine clearance at T0 and T1;
  * Liver enzymes at T0 and T1: alanine aminotransferase (ALT) and aspartate aminotransferase (AST);
  * T0 and T1 lipid profile: low density lipoproteins (LDL-c) and triglycerides (TG);
  * Complications of type 2 diabetes;
  * Treatment of cancer;
  * Family history of cancer.

SUMMARY:
Recent research has highlighted the significant relationship between type 2 diabetes mellitus and cancer, both prevalent and impactful on global health. The intrinsic correlation arises from shared metabolic processes, particularly a systemic and chronic inflammatory state driven by factors like obesity, dyslipidemia, and hyperglycemia. This leads to the creation of a self-sustaining microenvironment known as meta-inflammation, promoting cancer development through DNA damage, oxidative stress, and the influence of hormones like leptin. The hyperglycemic environment in diabetes contributes to cancer development, supporting the Warburg effect and insulin-related mechanisms. This study aims to identify risk factors associated with diabetes that impact tumor development and progression, crucial for guiding effective preventive strategies in clinical practice.

Primary objective of the study:

- identify the risk factors affecting the occurrence of cancer in the population affected by type 2 diabetes mellitus;

Secondary objectives of the study:

* description of the demographic, clinical and first-line therapy characteristics of patients diagnosed with type 2 diabetes mellitus;
* assess risk factors for recurrence, presence of a second tumour not related to the first and the presence of both events in patients who have had a tumor within 10 years of diagnosis of diabetes;
* assess the relationship between the characteristics of patients and the time to the onset of cancer.

DETAILED DESCRIPTION:
Study design This study is a monocentric retrospective cohort study based on the data available in the Smart Digital Clinic (Meteda Srl) electronic medical record.

Participating centre Surgery of Endocrinology and Diabetology of the SCDU of Novara, University of Eastern Piedmont. Responsible: Prof.ssa Flavia Prodam

Subjects Will be included in the study all patients visited at the Endocrinology and Diabetology surgery of the AOU Major of the Charity of Novara for an initial diagnosis of diabetes mellitus type 2 between 1990 and 2010.

Inclusion criteria

* Legal age
* Diagnosis of type 2 diabetes mellitus Exclusion criteria
* Diagnosis of cancer before diagnosis of type 2 diabetes
* Diagnosis of diabetes secondary to other diseases
* Diagnosis of diabetes secondary to other drugs
* Diagnosis of diabetes following surgery

Duration of study: 24 months

Follow-up and events of interest Patients included in the study will be followed from the date of diagnosis of type 2 diabetes mellitus until the date of the last available examination.

During the follow-up, for all patients included, the year of onset of the first cancer after the diagnosis of diabetes and the type of tumor will be detected. From this information it will be possible to calculate the time between the diagnosis of diabetes and the onset of cancer (measured in years).

For patients who have developed a first tumor will also be detected:

1. Recurrence of cancer (year of onset of recurrence)
2. Diagnosis of second tumour not related to primary tumour (year of onset, type of tumour) The diagnosis of cancer will be identified through the extraction system from the electronic medical record Smart Digital Clinic (Meteda Srl), using key words relevant to the area of cancer, identified in the section of the medical history. The key words will be: metastasis, adenocarcinoma, carcinoma, neoplasm, secondary/s, sarcoma, tumor, adenoma, lymphoma, leukemia, glioma, glioblastoma, ependymoma, basalioma, epithelium, melanoma, mesothelioma, cordoma, anaplastic, differentiated, undifferentiated, meningioma, multiple myeloma, small cell carcinoma, timoma, craniopharyngioma, neuroendocrine, LH, LNH, K, GIST, HCC and NET.

Data collection

For each patient, the following variables will be extracted from the Smart Digital Clinic electronic medical record for all visits available after diagnosis, where possible:

* Gender and age;
* Smoking habits and alcohol consumption (units per day);
* Weight and body mass index (BMI) at first (T0) and last visit (T1);
* Given by the diagnosis of type 2 diabetes mellitus;
* Treatment of type 2 diabetes mellitus at T0 and T1;
* Levels of glycated hemoglobin (hba1c) at T0 and T1, mean hba1c and mean fasting blood sugar;
* Creatinine clearance at T0 and T1;
* Liver enzymes at T0 and T1: alanine aminotransferase (ALT) and aspartate aminotransferase (AST);
* T0 and T1 lipid profile: low density lipoproteins (LDL-c) and triglycerides (TG);
* Complications of type 2 diabetes mellitus;
* Treatment of cancer;
* Family history of cancer; The diagnosis of type 2 diabetes mellitus is confirmed at diabetological centres or, in some cases, by general practitioners who refer patients to specialised diabetological centres. The accuracy of the diagnosis will be confirmed by crossing the Piedmont Diabetic Registry (PDR) and involving a second person to ensure a precise assessment.

BMI categories will be divided into underweight (BMI <18.5 Kg/m2), normal weight (BMI 18.5 - 25 Kg/m2), and overweight (BMI >25 Kg/m2).

With regard to the treatment of type 2 diabetes mellitus, participants will be categorised and grouped for statistical purposes in the following classes:

* Dietary therapy;
* Metformin/Acarbosio;
* Sulfanilurea;
* Metformin + GLP1/ DDPIV inhibitors (DDPIVi) or only GLP1 or only DDPIVi;
* Metformin + SGLT2i inhibitors (SGLT2i) or only SGLT2i;
* Basal insulin + GLP1/DDPIVi +/- Metformin;
* Basal insulin +/- Metformin +/- SGLT2i;
* Insulin basal bolus;
* Basal insulin bolus +/- Metformin +/- SGLT2i. In addition, complications of metabolic pathology will be extracted from the dedicated section of the program, where are systematically recorded and organized, and the diagnosis of which is conducted in accordance with the appropriate guidelines. These complications will be divided into the following categories: vasculopathy, neuropathy, hypertension, heart disease, kidney failure and retinopathy.

Finally, as regards cancer pathology, a categorization of treatment will be carried out in three classes: chemotherapy, surgery and radiation therapy.

In addition, the types of cancer will be divided in order to ensure greater homogeneity between groups, including the nervous system, head and neck, thorax, gastrointestinal, gynecological, urinary tract, male genital system, skin, blood, breast, soft tissues, endocrine glands and neuroendocrine tumors. This information will be collected at the diabetes diagnosis visit and at the last visit before the onset of cancer for the subjects experiencing the event and at the last available visit for the remaining subjects.

EXPECTED RESULTS Through this research, the investigators aim to obtain new information on the study population in order to better understand the possible correlation between the two pathologies. This will allow us to identify the risk factors associated with metabolic pathology that can affect the development time of cancer pathologies, as well as to identify those that could contribute to carcinogenesis itself.

This knowledge will allow us to define the role of hyperglycemia, obesity and other factors or behaviors at risk in the field of cancer in order to act with appropriate prevention strategies, thus considering the tumor pathology as one of the possible complications of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Legal age
* Diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

* Diagnosis of cancer before diagnosis of type 2 diabetes
* Diagnosis of diabetes secondary to other diseases
* Diagnosis of diabetes secondary to other drugs
* Diagnosis of diabetes following surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 779 patients with diabetes mellitus type 2 and with at least 18 years old.
Sampling Method: Probability Sample
Enrollment: 779 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-02-04 (Estimated); Study Completion 2025-02-04 (Estimated)

PRIMARY OUTCOMES:
Smoking assessment at first visit | Assessment of data at time 0 (first clinical visit)
  identify the risk factors affecting the occurrence of cancer in the population affected by type 2 diabetes mellitus: During the first examination, the history of each patient was investigated, evaluating whether they were smokers, non-smokers or ex smokers
Alcool consumption at first visit | Assessment of data at time 0 (first clinical visit)
  identify the risk factors influencing the onset of cancer in the population affected by type 2 diabetes mellitus: During the first examination, the history of each patient was studied, assessing whether I consume alcohol and in what amount. <1 alcohol unit or greater than 2 alcohol units were used as cutoffs to subdivide the patients considered.
BMI assessment at first visit | Assessment of data at time 0 (first clinical visit)
  identify the risk factors influencing the onset of cancer in the population affected by type 2 diabetes mellitus: During the first examination, the history of each patient was studied, measuring weight and height to calculate the BMI of each patient. The ranges considered are: underweight <18.5, normal weight 18.5-25 and overweight >25.
Glycated assessment at first visit | Assessment of data at time 0 (first clinical visit)
  identify the risk factors influencing the onset of cancer in the population affected by type 2 diabetes mellitus: During the first examination, the history of each patient was studied, measuring the glycate of each patient. The considered cutoff is < or equal to 8%, where 8% is the limit for glycemic decompensation.

SECONDARY OUTCOMES:
First-line therapy characteristics assessment at first visit | Assessment of data at time 0 (first clinical visit)
  Detection of drug therapy given at the first visit considering the medical record. The therapies considered were: Dietotherapy, Metformin/Acarbosio, Sulfanilurea, Metformin + GLP1/DDPIVi or GLP1 alone or DDDPIVi alone, Metformin + SGLT2i or SGLT2i alone, Basal insulin + GLP1/DPIVi +/- Metformin, Basal Insulin +/- Metformin + SGT2i, Insulin Basal Bolus, Insulin Basal Bolus +/- Metformin +/- SGLT2i
Primary outcomes and recurrence or presence of a secondary tumor | Assessment of data at time 0 (first clinical visit)
  Considering the risk factors measured as primary findings, it was intended to observe a possible association with those who had recurrence or with the development of a secondary tumour unrelated to the first, within 10 years of the diagnosis of diabetes. Detected during first clinical visit signed in the medical record
Relationship between patients characteristics and the time onset of cancer considering anthropometric and biochemical data | Assessment of data at time 0 (first clinical visit)
  Assess the relationship between the characteristics of patients and the time to the onset of cancer using medical record
Tumour characterization in the considered population, detected at the first clinical visit | Assessment of data at time 0 (first clinical visit)
  Characterization of tumors: tumors of the nervous system, head neck, thoracic, gastrointestinal, gynecological, urological, male genital, cutaneous, haematological, breast, soft tissue, endocrine glands, neuroendocrine and bone tumors. Detected during first clinical visit considering the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Prodam, MD PhD, Principal Investigator — AOU Maggiore della Carità di Novara
Locations (1):
- SCDU Endocrinology, AOU Ospedale Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fu Z, Gilbert ER, Liu D. Regulation of insulin synthesis and secretion and pancreatic Beta-cell dysfunction in diabetes. Curr Diabetes Rev. 2013 Jan 1;9(1):25-53. PMID 22974359
- [Background] Rojas A, Schneider I, Lindner C, Gonzalez I, Morales MA. Association between diabetes and cancer. Current mechanistic insights into the association and future challenges. Mol Cell Biochem. 2023 Aug;478(8):1743-1758. doi: 10.1007/s11010-022-04630-x. Epub 2022 Dec 24. PMID 36565361
- [Background] Cignarelli A, Genchi VA, Caruso I, Natalicchio A, Perrini S, Laviola L, Giorgino F. Diabetes and cancer: Pathophysiological fundamentals of a 'dangerous affair'. Diabetes Res Clin Pract. 2018 Sep;143:378-388. doi: 10.1016/j.diabres.2018.04.002. Epub 2018 Apr 19. PMID 29679627
- [Background] Francisco V, Pino J, Campos-Cabaleiro V, Ruiz-Fernandez C, Mera A, Gonzalez-Gay MA, Gomez R, Gualillo O. Obesity, Fat Mass and Immune System: Role for Leptin. Front Physiol. 2018 Jun 1;9:640. doi: 10.3389/fphys.2018.00640. eCollection 2018. PMID 29910742
- [Background] Chiefari E, Mirabelli M, La Vignera S, Tanyolac S, Foti DP, Aversa A, Brunetti A. Insulin Resistance and Cancer: In Search for a Causal Link. Int J Mol Sci. 2021 Oct 15;22(20):11137. doi: 10.3390/ijms222011137. PMID 34681797
- [Background] Yakar S, Leroith D, Brodt P. The role of the growth hormone/insulin-like growth factor axis in tumor growth and progression: Lessons from animal models. Cytokine Growth Factor Rev. 2005 Aug-Oct;16(4-5):407-20. doi: 10.1016/j.cytogfr.2005.01.010. PMID 15886048
- [Background] Mao Z, Zhang W. Role of mTOR in Glucose and Lipid Metabolism. Int J Mol Sci. 2018 Jul 13;19(7):2043. doi: 10.3390/ijms19072043. PMID 30011848
- [Background] Saxton RA, Sabatini DM. mTOR Signaling in Growth, Metabolism, and Disease. Cell. 2017 Mar 9;168(6):960-976. doi: 10.1016/j.cell.2017.02.004. PMID 28283069
- [Background] Laplante M, Sabatini DM. mTOR signaling in growth control and disease. Cell. 2012 Apr 13;149(2):274-93. doi: 10.1016/j.cell.2012.03.017. PMID 22500797
- [Background] Shlomai G, Neel B, LeRoith D, Gallagher EJ. Type 2 Diabetes Mellitus and Cancer: The Role of Pharmacotherapy. J Clin Oncol. 2016 Dec 10;34(35):4261-4269. doi: 10.1200/JCO.2016.67.4044. Epub 2016 Nov 7. PMID 27903154
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT06299800/Prot_SAP_000.pdf